## **COVER PAGE**

<u>Title</u>: Minimally invasive detection of sleep apnoea and effects of nCPAP therapy: a proof-of-concept study.

**NCT**: not available

<u>Date of the document (most recent update):</u> October 22, 2018.

# **CLINICAL PROJECT FOND ERASME 2018-19**

## Minimally invasive detection of sleep apnoea and effects of nCPAP therapy: a proof-of-concept study

**Department of Cardiology** 

and

**Sleep Laboratory** 

Hôpital Erasme

**Bruxelles** 

**Belgium** 

### 1. Background

Basic concepts: from anatomic architecture to ventricular function

According with the model of a helical myocardium, described for the first time by Turrent and Guasp in the 1954 (1), cardiomyocytes are functionally divided in an upper-basal loop, where they are disposed circumferentially, and in an apical-loop where they are arranged in a right-handed and left-handed helices to form a vortex at the apex. This figure-8 configuration, along with interactions between cardiomyocytes, is responsible for the complex beat-to-beat mechanical motion of the heart: a global counter-clockwise twist during the pre-ejection phase, a vigorous counter-clockwise apical twist during ejection and a clockwise apical untwist during the isovolumic phase (2), in order to boost the blood mass into the main vasculature with a helical mouvement. Changes in LV pre-load, after-load (3) and contractility (3-5) affect LV twist mechanics.

Recording the beat-to-beat blood velocity and heart-induced chest wall motions: ballistocardiography and seismocardiography

In the late 1887, Gordon assumed that the body moves with each heart beat (6). Nowadays, we can confirm Gordon's hypothesis and state that the micro-movements of the body are due to the blood ejection velocity into the ascending aorta (7, 8). These "cardiogenic body movements" can be measured by the mean of ballistocardiography (BCG), which measures the displacement, velocity and acceleration of the body in response to the displacements of the heart and blood in the main vasculature (9); and the seismocardiography (SCG) which assesses the micro-vibrations produced by the heart contraction and blood ejection into the vascular tree which are transmitted to wall chest, where they are recorded (10).

Because of the advent of more performant imaging technologies, such as bi-dimensional and tri-dimensional echocardiography and cardiac resonance, BCG and SCG are not used anymore nowadays (11).

Experimental application of BCG and SCG

A large body of studies exists on the potential applicability of BCG and SCG in clinical practice. For instance, SCG records changes in the ventricular wall motion and compliance after an ischaemic event to a similar extent than an ECG (12), and when combined with an ECG, the accuracy of detecting physiologically significant coronary artery disease is greater than with an ECG recording alone (13). BCG was successfully used in automatic detection of atrial fibrillation (14), and to predict adverse clinical outcome in patients with heart failure (15).

Apart from the clinical setting, BCG and SCG have been used to analyse cardiac function in a microgravity environment. The first 3D-BCG recordings were made during the 4<sup>th</sup> expedition on the Saluyt-6 orbital station by the Soviets (16), as well as during the Spacelab mission in 1993 (17). 3D- BCG was also used to assess cardiac function (pre-ejection period (PEP)) and left ventricular ejection time (LVET)) on 5 healthy volunteers during the European Space Agency parabolic flight campaigns (18).

SCG and BCG signals: from parameters recording to biological interpretation

The SCG records the base-to-apex rotational movements transferred to the chest wall in the form of microvibrations. Several parameters of biological interest can be derived from SCG signals, especially the amplitude and temporal signals. The amplitude signals are related to left ventricular pressure (19), stroke volume and aortic blood pressure (20). Temporal signals provide information about ventricular function: namely a) PEP, a marker of cardiac contractility, b) LVET, c) the PEP/LVET ratio, a heart rate independent parameter and d) the isovolumic relaxation time (IVRT), which reflects the cardiac performance during the diastolic phase of the cardiac cycle (21). The BCG records also several waveforms, three of which are likely

of main importance for sleep apnoea monitoring: namely the "I", "J" and "K" waves (7, 8). These waves are elicited by the ventricular contraction which occurs after the QRS complex on the ECG. They represent the body movements in response to the cardiac blood ejection (22). Should the thoracic aorta be simplified into an ascending and a descending tube, on whom blood pressure and volume flow rate forces act in opposite directions, then the BCG waveforms represents the sum of those forces (8). Various cardiovascular parameters can be estimated from the BCG signal, and are shortly presented below. The J wave of the BCG represents the point of highest amplitude in the BCG waveform; heart rate can be determined by the time interval between consecutive J peaks, the J-J intervals (23). Various algorithms can assess heart rate from BCG signals (24-28). Also, heart rate variability, a non-invasive tool to assess cardiac sympathetic and parasympathetic modulation (29), can be calculated from BCG peak intervals, without the need of RR interval calculations obtained from ECG recordings. Changes in BCG waveforms amplitude are related to stroke volume (SV) and cardiac output (CO) modifications in healthy subjects (30, 31). Finally, similarly to SCG, BCG measurements provide an estimation of the PEP (32, 33), and the LVET which indicates the percentage of the cardiac cycle devoted to ejection as compared to ventricular filling (34, 35).

Sleep disordered breathing and their cardiovascular impact: why detect them?

Sleep apnoea syndrome is a common chronic respiratory disease characterised by cyclic airflow cessations during sleep. Clinically, they are classified in three entities; obstructive, where the airflow cessation is due to upper airways collapse; central, where the airflow cessation arise from a central lack in driving to the breathing muscles with no compensatory respiratory efforts; mixed, characterised by an initial central event followed by an obstructive one. Nowadays, up to 24% of men and to 9% of women aged 30 to 60 years disclose already an asymptomatic and underdiagnosed sleep disorder breathing (SDB) (36). Its current high prevalence will supposedly increase in the future years, as a result of the obesity pandemic in an ageing population. SDB is a potential cardiovascular risk factor (37). A patent causal relationship between SDB and cardiovascular disease has not been clearly established until now, but several chronic patho-physiological mechanisms could make sense in supporting such a link. Intermittent hypoxaemia, due to cycled upper airway collapse, is responsible for abnormal sympathetic activation (38), endothelial dysfunction (39), oxidative stress (40) and inflammation (41), all of which are related to cardiovascular illnesses, especially hypertension (42), atherosclerosis (43), cardiac arrhythmias (44), heart failure (45), and coronary artery disease (46). SDB is, likewise, positively correlated with an increased morbidity and mortality in the cardiovascular population (47, 48) and seems to be an independent predictive factor in cardiovascular mortality after an acute coronary syndrome (49).

Moreover, the classical profile of patients at risk of having SDB (obese subjects, Pickwickian syndrome) has changed in the past year, so that there are new categories of patients who should be evaluated for sleep apnoea, above all those with cardiovascular co-morbidities (50).

Sleep disordered breathing and kino-cardiography: a new and promising tool for unobstrusive recording of SDB and its impact on the cardiovascular system.

Complete laboratory polysomnography (PSG) is the gold standard to diagnose SDB (50, 51). However, it is an expensive, time-consuming and uncomfortable tool, limiting its wide-spread use despite the high frequency of SDB in the general population. However, considering the high prevalence of SDB in the general population and the change in the profile of patients at risk of SDB and then, who should be evaluated for, there is growing interest in the research of alternative strategies to reach the most of patients at possible. A number of home sleep testing devices has been proposed over years to screen patient at risk of SDB, but according to the guidelines, they are NOT recommended for patients with cardiovascular comorbidities (50). Moreover, the devices available nowadays do not provide any information on the direct impact of the apnoea on the cardiovascular system.

Nevertheless, taking into account the high prevalence of SDB and the limited accessibility of expensive sleep testing *on one side* and, *on the other side*, the marked recent technological advances in SCG and BCG technologies *as well as* the peculiar hemodynamic characteristics of sleep apnoea episodes, we wish to test

the hypothesis that modern SCG and BCG recordings can provide an highly accurate assessment of sleep apnoea, and evaluate the effects of nCPAP therapy.

There are several reasons to believe that the implementation of recent improvements in SCG-BCG will allow a precise quantification of such sleep-related events:

- 1) The cyclic pharynx collapses during sleep are associated to brain arousal, intrathoracic pressure swings (the so called 'Mueller manoeuvres'), and intermittent episodes of hypoxaemia and reoxygenation (45). When respiration resumes, the cardiac output faces a markedly increased peripheral sympathetic activity, leading to sudden rises in systemic blood pressure, and reflex reductions in heart rate, while the opposite occurs during the periods of respiratory collapse. As explained above, these changes are likely to induce marked modifications in the amplitude and temporal recording assessed by SCG recordings, as well as in the "I", "J" and "K" waves obtained from the BCG.
- 2) Previous studies which tested if BCG can detect sleep disturbances are encouraging, despite using remote techniques: Da Woon et al. used an unobtrusive polyvinylidene fluoride film sensor on a bed mattress to record BCG signals in a selected group of 10 OSA patients and 10 controls (52, 53). They calculated heart rate (HR) and heart rate variability (HRV) from J-J BCG interval and detected awakening periods in OSA patients with an accuracy of 97%. *The authors could however not determine why sleep was fragmented with this technique*. Zaho et al. also used a micro-movement sensitive bed mattress in subjects with a BMI < 35 kg/m² and no other concomitant cardiorespiratory disease (54). HRV was also retrieved from J-J BCG interval. However, *only selected periods of sleep were analysed for sleep-breathing events, a surrogate marker for obstructive, but not central apnoea*. Detection of these events was nevertheless achieved with a sensitivity of 98%, a specificity of 94%, and an accuracy of 98% (55). Last, Dehkordi et al. showed that it was possible to distinguish between central and obstructive events by recording acceleration from the suprasternal notch, the thorax and the abdomen (56). The subjects investigated were however *only normal volunteers* who performed several voluntary breaths hold in the presence of an oral nasal flow detector.
- 3) The unique expertise of our research team is that we are capable to record SCG and BCG signals in 3 dimensions (57, 58), both linearly and rotationally (16-18). While the above mentioned studies (52-56) assessed BCG changes only in a horizontal plane (x and y axis), which is not representative of the complex cardiac mechanic, we are capable to record these changes in a third anteroposterior dimensions (z axis). This is important because of the anterior-posterior direction of the aortic arch. In addition, as emphasized in the introduction of this research proposal, an important component of the body reaction to the heart movements is rotational, which we are capable to record in 3 dimensions. Overall the combined SCG and BCG 3D-linear and 3D-rotational signals represent 6 degrees of freedom (DOF) while past BCG had only 2-DOF. For simplicity, this 6 DOF signal combination will be designated as Kino-cardiography (KCG) recordings in this research proposal. We anticipate that the unique KCG properties will considerably increase our detection capability of obstructive and central apnoea, as compared to previous studies.

### 2. Aims and hypothesis tested

The main hypothesis tested in our study is that KCG provides sensitive and accurate measures of obstructive and central apnoea as compared to state-of-the-art polysomnography. Our secondary hypotheses are related to modifications in the SCG and BCG parameters during the apnoea and the effects of nCPAP therapy: we believe that the KCG signals are profoundly affected by the apnoea and they are reversed to the normal baseline with the CPAP. These hypotheses will be tested through a series of studies in normal volunteers and patients.

#### 1-MAIN HYPOTHESES:

<u>Group A.</u> After a fine tuning period of the KCG signal post processing to maximise the sensitivity and specificity of voluntary apnoea detection in health subjects, we will start the first validation study. In 46 healthy volunteers, a computer program will generate random instructions of periods of normal breathing, voluntary end-expiratory breathing cessations periods (as surrogate of central apnoea) and Muller's manœuvre (as surrogate of obstructive apnoea). Meanwhile, the KCG will record the above-mentioned parameters. The number and duration of voluntary central and obstructive apnoea will be assessed in the KCG recordings, not knowing how many were actually generated by the computer program. We will also record the ECG, heart rate, beat to beat non-invasive blood pressure (Finometer), humeral blood pressure (Dinamap), ventilation, end-tidal  $CO_2$  (AD instruments),  $O_2$  saturation (Nellcor), cardiac output (CO) (Philips).

**Group B.** In patients suspected of sleep apnoea and admitted to the sleep unit of the Erasme hospital to perform sleep test as required by their medical condition, we will simultaneously record KCG and PSG and qualitatively compare the data. Bland-Altman plots will analyse the agreement between the sleep recordings obtained with the two methods. Peculiar attention will be paid to the accuracy of the detection of obstructive *versus* central *versus* mixed apnoea, of awakenings, and of the time spend in bed. In this second phase of the study, we plan to record these parameters only in selected patients, who will not disclose marked abnormalities which could hamper the reliability of the KCG recordings, namely moderate or severe valvular disease, permanent atrial fibrillation or frequent premature contractions, atrio-ventricular conduction disturbances, medications which reduce heart rate and heart rate variability (beta blockers, anti-arrhythmic drugs, calcium blockers, ...), cardiac rhythm driven by a pace maker, heart failure of any origin, neurological diseases responsible for abnormal movements (restless leg syndrome, Parkinson disease, ataxia ...).

**Group C**. In patients with a diagnosis of OSA, we will determine if KCG is capable to reliably assess the efficacy of the nCPAP therapy in comparison to simultaneous PSG recording. Ongoing adjustment in CPAP therapy pressure during the night, and its effect on cardiovascular haemodynamic assessed by the KCG, will be taken into account as well. The capability of the technique to detect changes in sleep quality will be tested both *within* subjects (before vs. after nCPAP therapy in the same patient) as well *among* the subjects investigated. The same restriction in the recruitment of the subjects of group B will be applied for the present group.

<u>Group D</u>. After validation of the three previous steps, we plan to extend the recordings on 100 unselected consecutive patients who will undergo PSG recordings because of complains of sleep apnoea. This will validate the clinical usefulness of KCG recording for the detection of sleep apnoea even in patients with multiples co-morbidities.

#### 2-SECONDARY HYPOTHESES

We will test the hypothesis that the apnoeic events profoundly affected the KCG signals (PEP, LVET and PEP/LVET ratios). These parameters are affected by changes in cardiac pre- and after- load and sympathetic activity on myocardial contractility. Similarly, we plan to test the hypothesis that the isovolumic relaxation time (IVRT), an index of diastolic performance during the cardiac cycle, will be altered during the obstructive apneas, because marked variation in intrathoracic pressure result in large increases in LV transmural gradient and thereby reduce LV compliance. CPAP therapy should markedly reduce the nighttime variability in these parameters.

We will also asses the R-J interval which is related to blood pressure and determine if this parameter rises during the apneas and arousals when sympathetic activity is increased. Determination of the J-J intervals and the corresponding HRV, which is under strong autonomic control, should also present distinct changes in OSA patients, as compared to subjects receiving efficacious nCPAP therapy.

Last, breathing effort variations will be assessed. This refers to the mechanical interaction between respiration and KCG signals when sleep apnea occurs, independently from an autonomic nervous modulation of heart rate variability: when the obstructive apneic event occurs, the airflow decreases, which result in a

breathing effort thereafter. We will test the hypothesis that theses respiratory abnormalities are readily detectable by the KCG.

#### 3. Methods

Study design and recruitment, expertise of the research group

Study A is an interventional pre-study on voluntary breath holding on healthy subjects. The parameter taken into consideration for sample size calculation in this group is the total (linear and rotational) systolic kinetic energy of the SCG (S\_sys\_kin) and the rolling ratio between the mean value and the standard deviation of this parameter:  $H = Mean(S_sys_kin) / Std(S_sys_kin)$ . H discriminated voluntary obstructive apneas from episodes of normal respiration in a healthy volunteer (H = 1.1627 and 0.2308, respectively). The sample size is determined according to:  $2 \cdot (Zalpha + Z1-beta)2 \cdot sigma2 / Delta2$ , where alpha = 5% is the accepted error, leading to Zalpha = 1.96 (2-sided); beta = 95% is the power of the study, leading to Z1-beta = 1.64; sigma is the estimated standard deviation of H; delta is the estimated effect of obstructive sleep apnea on H in patients. Sigma (Hbaseline) = 0.1247 was obtained by H determinations on a group of healthy subjects who were breathing regularly. The difference in H during regular breathing and voluntary obstructive apnea, divided by 10 (because voluntary apneas may have induced larger changes than those experienced by patients) is Delta = (1.1627 - 0.2308) / 10 = 0.09319. Thus, the estimated sample size for study A is 46.

Studies B and C are observational investigations on subjects referred for PSG as required by their medical condition and which fulfill the inclusion/exclusion criteria described previously. The number of subjects will be calculated accordingly to the results of the pre-study (group A).

Study D is an observational prospective investigation conducted on unselected consecutive patients without recruitment restrictions, in order to validate the KCG on the real population. Since we do not know how many patients will be necessary for the validation of our screening device, we speculate a size simple of 100 subjects.

Because the KCG device is not intrusive, we do not anticipate difficulties in the recruitment. Our study will not affect in any manner the regular medical care of the patients admitted to the sleep laboratory. The present research proposal is in line with my promotor's expertise, P. van de Borne, P-F. Migeotte and G. Loas, in the study of sleep physiology (59-63), and sleep apnea (60, 61):

## 4. Perspectives

As explained above, SDB is a widespread disease with detrimental health effects and its prevalence is supposed to increase in the future years, as the result of the obesity pandemic in an ageing population. PSG is the gold standard for the diagnosis of sleep related disorders but it is an expensive, uncomfortable and time-consuming tool, limiting its use in the daily clinical practice, despite the high prevalence of SDB. Several home sleep tests have been proposed to screen patients suspected for SDB, but they disclose several limitations and are not recommended for patients with cardiovascular, respiratory, metabolic or neurologic co-morbidities (50). We strongly believe that the less cumbersome (57-60) KCG will screen patients for SDB accurately. One of its unique features (57-60) is also that it can directly identify the consequences of SDB and nCPAP therapy on the cardiovascular system, and in especially the presence of frequently associated cardiac arrhythmias (44). With a more efficient pre-screening, those who are most likely to be eligible for nCPAP therapy will have a better access to the currently existing sleep laboratory facilities. To summarize, we aim 1) to propose a new screening tool for patients at risk of SDB, 2) to stratify patients with SDB for adverse cardiovascular events, and 3) to highlight new physio-pathological aspect of sleep apnoea. The present research project has thus the potential of improving sleep apnoea patients care and health, at no additional societal costs.

#### 5. References

- 1. Kocica MJ, Corno AF, Lackovic V, Kanjuh VI. The helical ventricular myocardial band of Torrent-Guasp. Seminars in thoracic and cardiovascular surgery Pediatric cardiac surgery annual. 2007:52-60.
- 2. Buckberg G, Hoffman JI, Mahajan A, Saleh S, Coghlan C. Cardiac mechanics revisited: the relationship of cardiac architecture to ventricular function. Circulation. 2008;118(24):2571-87.
- 3. Dong SJ, Hees PS, Huang WM, Buffer SA, Jr., Weiss JL, Shapiro EP. Independent effects of preload, afterload, and contractility on left ventricular torsion. The American journal of physiology. 1999;277(3 Pt 2):H1053-60.
- 4. Hansen DE, Daughters GT, 2nd, Alderman EL, Ingels NB, Stinson EB, Miller DC. Effect of volume loading, pressure loading, and inotropic stimulation on left ventricular torsion in humans. Circulation. 1991;83(4):1315-26.
- 5. Stohr EJ, Shave RE, Baggish AL, Weiner RB. Left ventricular twist mechanics in the context of normal physiology and cardiovascular disease: a review of studies using speckle tracking echocardiography. Am J Physiol Heart Circ Physiol. 2016;311(3):H633-44.
- 6. Gordon JW. Certain Molar Movements of the Human Body produced by the Circulation of the Blood. Journal of anatomy and physiology. 1877;11(Pt 3):533-6.
- 7. Jafari Tadi M, Lehtonen E, Saraste A, Tuominen J, Koskinen J, Teras M, et al. Gyrocardiography: A New Non-invasive Monitoring Method for the Assessment of Cardiac Mechanics and the Estimation of Hemodynamic Variables. Sci Rep. 2017;7(1):6823.
- 8. Kim CS, Ober SL, McMurtry MS, Finegan BA, Inan OT, Mukkamala R, et al. Ballistocardiogram: Mechanism and Potential for Unobtrusive Cardiovascular Health Monitoring. Sci Rep. 2016;6:31297.
- 9. Wiard RM, Kim HJ, Figueroa C, Kovacs GT, Taylor CA, Giovangrandi L. Estimation of central aortic forces in the ballistocardiogram under rest and exercise conditions. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2009;2009:2831-4.
- 10. Bozhenko BS. [Seismocardiography--a new method in the study of functional conditions of the heart]. Terapevticheskii arkhiv. 1961;33:55-64.
- 11. Giovangrandi L, Inan OT, Wiard RM, Etemadi M, Kovacs GT. Ballistocardiography--a method worth revisiting. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2011;2011:4279-82.
- 12. Salerno DM, Zanetti JM, Green LA, Mooney MR, Madison JD, Van Tassel RA. Seismocardiographic changes associated with obstruction of coronary blood flow during balloon angioplasty. Am J Cardiol. 1991;68(2):201-7.
- 13. Wilson RA, Bamrah VS, Lindsay J, Jr., Schwaiger M, Morganroth J. Diagnostic accuracy of seismocardiography compared with electrocardiography for the anatomic and physiologic diagnosis of coronary artery disease during exercise testing. Am J Cardiol. 1993;71(7):536-45.
- 14. Brueser C, Diesel J, Zink MD, Winter S, Schauerte P, Leonhardt S. Automatic detection of atrial fibrillation in cardiac vibration signals. IEEE journal of biomedical and health informatics. 2013;17(1):162-71.
- 15. Giovangrandi L, Inan OT, Banerjee D, Kovacs GT. Preliminary results from BCG and ECG measurements in the heart failure clinic. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2012;2012:3780-3.
- 16. Baevskii RM, Funtova, II. [Ballistocardiographic studies during the 4th expedition on the Saliut-6 orbital station]. Kosm Biol Aviakosm Med. 1982;16(5):34-7.
- 17. Prisk GK, Verhaeghe S, Padeken D, Hamacher H, Paiva M. Three-dimensional ballistocardiography and respiratory motion in sustained microgravity. Aviation, space, and environmental medicine. 2001;72(12):1067-74.
- 18. Migeotte PF, Deliere Q, Tank J, Funtova I, Baevsky R, Neyt X, et al. 3D-ballistocardiography in microgravity: comparison with ground based recordings. Conference proceedings: Annual International

Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2013;2013:7012-6.

- 19. Gemignani V, Bianchini E, Faita F, Lionetti V, Campan M, Recchia FA, et al. Transthoracic sensor for noninvasive assessment of left ventricular contractility: validation in a minipig model of chronic heart failure. Pacing and clinical electrophysiology: PACE. 2010;33(7):795-803.
- 20. Bombardini T, Gemignani V, Bianchini E, Venneri L, Petersen C, Pasanisi E, et al. Arterial pressure changes monitoring with a new precordial noninvasive sensor. Cardiovascular ultrasound. 2008;6:41.
- 21. Di Rienzo M, Vaini E, Castiglioni P, Merati G, Meriggi P, Parati G, et al. Wearable seismocardiography: towards a beat-by-beat assessment of cardiac mechanics in ambulant subjects. Autonomic neuroscience: basic & clinical. 2013;178(1-2):50-9.
- 22. Inan OT, Etemadi M, Wiard RM, Kovacs GT, Giovangrandi L. Novel methods for estimating the ballistocardiogram signal using a simultaneously acquired electrocardiogram. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2009;2009:5344-47.
- 23. Inan OT, Migeotte PF, Park KS, Etemadi M, Tavakolian K, Casanella R, et al. Ballistocardiography and seismocardiography: a review of recent advances. IEEE journal of biomedical and health informatics. 2015;19(4):1414-27.
- 24. Choi BH, Chung GS, Lee JS, Jeong DU, Park KS. Slow-wave sleep estimation on a load-cell-installed bed: a non-constrained method. Physiological measurement. 2009;30(11):1163-70.
- 25. Jansen BH, Larson BH, Shankar K. Monitoring of the ballistocardiogram with the static charge sensitive bed. IEEE Trans Biomed Eng. 1991;38(8):748-51.
- 26. Shin JH, Choi BH, Lim YG, Jeong DU, Park KS. Automatic ballistocardiogram (BCG) beat detection using a template matching approach. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2008;2008:1144-6.
- 27. Bruser C, Winter S, Leonhardt S. Robust inter-beat interval estimation in cardiac vibration signals. Physiological measurement. 2013;34(2):123-38.
- 28. Paalasmaa J, Toivonen H, Partinen M. Adaptive Heartbeat Modeling for Beat-to-Beat Heart Rate Measurement in Ballistocardiograms. IEEE journal of biomedical and health informatics. 2015;19(6):1945-52.
- 29. Bisogni V, Pengo MF, Maiolino G, Rossi GP. The sympathetic nervous system and catecholamines metabolism in obstructive sleep apnoea. Journal of thoracic disease. 2016;8(2):243-54.
- 30. Castiglioni P, Faini A, Parati G, Di Rienzo M. Wearable seismocardiography. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2007;2007:3954-7.
- 31. Inan OT, Etemadi M, Paloma A, Giovangrandi L, Kovacs GT. Non-invasive cardiac output trending during exercise recovery on a bathroom-scale-based ballistocardiograph. Physiological measurement. 2009;30(3):261-74.
- 32. Da He D, Winokur ES, Sodini CG. A continuous, wearable, and wireless heart monitor using head ballistocardiogram (BCG) and head electrocardiogram (ECG). Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2011;2011:4729-32.
- 33. Etemadi M, Inan OT, Giovangrandi L, Kovacs GT. Rapid assessment of cardiac contractility on a home bathroom scale. IEEE transactions on information technology in biomedicine: a publication of the IEEE Engineering in Medicine and Biology Society. 2011;15(6):864-9.
- 34. Di Rienzo M, Vaini E, Castiglioni P, Meriggi P, Rizzo F. Beat-to-beat estimation of LVET and QS2 indices of cardiac mechanics from wearable seismocardiography in ambulant subjects. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2013;2013:7017-20.
- 35. Ngai B, Tavakolian K, Akhbardeh A, Blaber AP, Kaminska B, Noordergraaf A. Comparative analysis of seismocardiogram waves with the ultra-low frequency ballistocardiogram. Conference proceedings:

Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2009;2009:2851-4.

- 36. Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993;328(17):1230-5.
- 37. Parish JM, Somers VK. Obstructive sleep apnea and cardiovascular disease. Mayo Clin Proc. 2004;79(8):1036-46.
- 38. Somers VK, Dyken ME, Clary MP, Abboud FM. Sympathetic neural mechanisms in obstructive sleep apnea. The Journal of clinical investigation. 1995;96(4):1897-904.
- 39. Belaidi E, Joyeux-Faure M, Ribuot C, Launois SH, Levy P, Godin-Ribuot D. Major role for hypoxia inducible factor-1 and the endothelin system in promoting myocardial infarction and hypertension in an animal model of obstructive sleep apnea. J Am Coll Cardiol. 2009;53(15):1309-17.
- 40. Lavie L. Oxidative stress in obstructive sleep apnea and intermittent hypoxia--revisited--the bad ugly and good: implications to the heart and brain. Sleep medicine reviews. 2015;20:27-45.
- 41. Shamsuzzaman AS, Winnicki M, Lanfranchi P, Wolk R, Kara T, Accurso V, et al. Elevated C-reactive protein in patients with obstructive sleep apnea. Circulation. 2002;105(21):2462-4.
- 42. Parati G, Lombardi C, Hedner J, Bonsignore MR, Grote L, Tkacova R, et al. Recommendations for the management of patients with obstructive sleep apnoea and hypertension. The European respiratory journal. 2013;41(3):523-38.
- 43. Hoyos CM, Melehan KL, Liu PY, Grunstein RR, Phillips CL. Does obstructive sleep apnea cause endothelial dysfunction? A critical review of the literature. Sleep medicine reviews. 2015;20:15-26.
- 44. Mehra R, Benjamin EJ, Shahar E, Gottlieb DJ, Nawabit R, Kirchner HL, et al. Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study. American journal of respiratory and critical care medicine. 2006;173(8):910-6.
- 45. Bradley TD, Floras JS. Sleep apnea and heart failure: Part I: obstructive sleep apnea. Circulation. 2003;107(12):1671-8.
- 46. Konecny T, Kuniyoshi FH, Orban M, Pressman GS, Kara T, Gami A, et al. Under-diagnosis of sleep apnea in patients after acute myocardial infarction. J Am Coll Cardiol. 2010;56(9):742-3.
- 47. Bradley TD, Floras JS. Obstructive sleep apnoea and its cardiovascular consequences. Lancet (London, England). 2009;373(9657):82-93.
- 48. Won CH, Chun HJ, Chandra SM, Sarinas PS, Chitkara RK, Heidenreich PA. Severe obstructive sleep apnea increases mortality in patients with ischemic heart disease and myocardial injury. Sleep Breath. 2013;17(1):85-91.
- 49. Milleron O, Pilliere R, Foucher A, de Roquefeuil F, Aegerter P, Jondeau G, et al. Benefits of obstructive sleep apnoea treatment in coronary artery disease: a long-term follow-up study. Eur Heart J. 2004;25(9):728-34.
- 50. [Recommendations for clinical practice. Obstructive sleep apnea hypopnea syndrome in adults]. Rev Mal Respir. 2010;27(7):806-33.
- 51. Fleetham J, Ayas N, Bradley D, Fitzpatrick M, Oliver TK, Morrison D, et al. Canadian Thoracic Society 2011 guideline update: diagnosis and treatment of sleep disordered breathing. Canadian respiratory journal. 2011;18(1):25-47.
- 52. Da Woon J, Su Hwan H, Hee Nam Y, Lee YJ, Do-Un J, Kwang Suk P. Nocturnal awakening and sleep efficiency estimation using unobtrusively measured ballistocardiogram. IEEE Trans Biomed Eng. 2014;61(1):131-8.
- 53. Park KS, Hwang SH, Jung DW, Yoon HN, Lee WK. Ballistocardiography for nonintrusive sleep structure estimation. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2014;2014:5184-7.
- 54. Weichao Z, Hongbo N, Xingshe Z, Yalong S, Tianben W. Identifying sleep apnea syndrome using heart rate and breathing effort variation analysis based on ballistocardiography. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2015;2015:4536-9.

- 55. Wang Z, Zhou X, Zhao W, Liu F, Ni H, Yu Z. Assessing the severity of sleep apnea syndrome based on ballistocardiogram. PLoS One. 2017;12(4):e0175351.
- 56. Dehkordi P, Marzencki M, Tavakolian K, Kaminska M, Kaminska B. Monitoring torso acceleration for estimating the respiratory flow and efforts for sleep apnea detection. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2012;2012:6345-8.
- 57. Lejeune L, Caiani EG, Prisk GK, Migeotte PF. Evaluation of ensemble averaging methods in 3D ballistocardiography. Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2014;2014:5176-9.
- 58. Migeotte PF, Lejeune L, Deliere Q, Caiani E, Casellato C, Tank J, et al. Three dimensional Ballistocardiogram and Seismocardiogram: what do they have in common? Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Annual Conference. 2014;2014:6085-8.
- 59. Dumont M, Jurysta F, Lanquart JP, Migeotte PF, van de Borne P, Linkowski P. Interdependency between heart rate variability and sleep EEG: linear/non-linear? Clinical neurophysiology: official journal of the International Federation of Clinical Neurophysiology. 2004;115(9):2031-40.
- 60. Janssen C, Pathak A, Grassi G, van de Borne P. Endothelin contributes to the blood pressure rise triggered by hypoxia in severe obstructive sleep apnea. Journal of hypertension. 2017;35(1):118-24.
- 61. Jurysta F, Lanquart JP, van de Borne P, Migeotte PF, Dumont M, Degaute JP, et al. The link between cardiac autonomic activity and sleep delta power is altered in men with sleep apnea-hypopnea syndrome. American journal of physiology Regulatory, integrative and comparative physiology. 2006;291(4):R1165-71.
- 62. Jurysta F, van de Borne P, Lanquart JP, Migeotte PF, Degaute JP, Dumont M, et al. Progressive aging does not alter the interaction between autonomic cardiac activity and delta EEG power. Clinical neurophysiology: official journal of the International Federation of Clinical Neurophysiology. 2005;116(4):871-7.
- 63. Jurysta F, van de Borne P, Migeotte PF, Dumont M, Lanquart JP, Degaute JP, et al. A study of the dynamic interactions between sleep EEG and heart rate variability in healthy young men. Clinical neurophysiology : official journal of the International Federation of Clinical Neurophysiology. 2003;114(11):2146-55.